CLINICAL TRIAL: NCT01914510
Title: Phase II Study of Oral ENMD-2076 Administered to Patients With Ovarian Clear Cell Carcinomas
Brief Title: A Study of ENMD-2076 in Ovarian Clear Cell Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENMD-2076-OCC
Record Dates: First submitted 2013-07-11; First posted 2013-08-02 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Ovarian Clear Cell Carcinoma
Keywords: ovarian; cancer; clear cell; ENMD-2076; oral; capsule
MeSH Terms: conditions — Neoplasms | interventions — ENMD 2076

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ENMD-2076 (Experimental): ENMD-2067 will be taken orally at a dose of 275 mg, once a day, everyday. Patients with a body surface area of less than 1.65 m2 will receive a starting dose of 250 mg, once a day, everyday.
  Interventions: Drug: ENMD-2076

INTERVENTIONS:
Drug: ENMD-2076

SUMMARY:
This is a phase 2 study to see how useful, safe, and tolerable an investigational drug called ENMD-2076 is in treating patients with ovarian clear cell carcinomas.

ENMD-2076 is an oral drug that works by blocking certain enzymes called Aurora A and tyrosine kinase from working. These enzymes are needed for cells to divide including cancer cells. ENMD-2076 also works by stopping the growth of new blood vessels which would provide the tumor with nutrients for it to grow. It is believed that by blocking Aurora A and tyrosine kinase enzymes from working and stopping new blood vessels from growing, the tumors may stop growing or shrink.

DETAILED DESCRIPTION:
During the study, participants will be asked to take ENMD-2076 once a day, everyday. Every 28 days will be called a cycle. While receiving the study drug, participants will be asked to visit the clinic for tests and procedures. During Cycle 1, participants will be asked to visit the clinic about once a week and during Cycle 2 and future cycles, participants will be asked to visit the clinic on days 1 and 15. As a part of the study, tumor tissue (archival and fresh tumor biopsy) will be taken for biomarker research. When participants stop the study drug, they will be asked to have an end of study drug visit.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically documented diagnosis of ovarian clear cell carcinoma.
* Any number of prior chemotherapy regimens will be allowed but must include 1 line of platinum based therapy, and may include chemotherapy, biologics or other targeted therapies (except for Aurora A targeted therapies).
* Meet RECIST criteria (version 1.1) within 28 days of start of treatment by having measurable disease defined as one or more lesions that can be accurately measured in one or more dimensions. Areas of previous radiation may not serve as measurable disease unless there is evidence of progression post radiation.
* At time of registration, if the patient has had previous treatment it must have been at least 4 weeks since major surgery or radiation therapy; four weeks from any other previous anti-cancer therapy including biologics. Patients must have recovered from their treatment-related events with the exception of alopecia.
* Are ≥18 years of age
* Have clinically acceptable laboratory screening results within certain limits specified below:

  * AST and ALT ≤ 2.5 times upper limit of normal (ULN) or less than or equal to 5 times ULN if liver metastases are present
  * Total bilirubin ≤ 1.5 x ULN
  * Creatinine ≤ 1.5 x UL
  * Absolute neutrophil count ≥ 1500 cells/mm
  * Platelets ≥ 150,000/mm3
  * Hemoglobin ≥ 9.0 g/dl
* Have an ECOG performance status of ≤ 2
* Women of child-producing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication. A serum pregnancy test within 72 hours prior to the initiation of therapy will be required for women of childbearing potential.
* Have the ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
* Able to tolerate oral medication.

Exclusion Criteria:

* Women who are pregnant or nursing
* Have active, acute, or chronic clinically significant infections or bleeding.
* Have uncontrolled hypertension (systolic blood pressure greater than 150mmHg or diastolic blood pressure greater than 100mmHg); or history of congestive heart failure (equal to or greater than Grade 2).
* Have active angina pectoris, stroke, previous myocardial infarction within the past 12 months and not clinically stable, or any other pre-existing uncontrolled cardiovascular condition.
* Have chronic atrial fibrillation or QTc interval corrected for heart rate of greater than 470 msec.
* Have additional uncontrolled serious medical or psychiatric illness.
* Require therapeutic doses of anti-coagulation with warfarin or other coumarin derivatives. However, treatment with low molecular weight heparin (LMWH) is allowed.
* Known CNS metastases
* Have any medical condition that would impair the administration of oral agents including recurrent bowel obstructions, inflammatory bowel disease or uncontrolled nausea, vomiting or diarrhea
* Have persistent 2+ protein by urinalysis (patients with 2+ proteinuria that have a spot protein:creatinine ratio of less than 0.3 may be enrolled) or a history of nephrotic syndrome
* Have an active or history of additional malignancy which in the opinion of the study doctor would make assessment of outcome difficult.
* Require treatment with drugs known to be potent inducers or inhibitors of CYP3A4 at the time of registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, Alberta
  - London Regional Cancer Program, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- ENMD-2076: ENMD-2067 will be taken orally at a dose of 275 mg, once a day, everyday, for the 28-day cycles. Patients with a body surface area of less than 1.65 m2 will receive a starting dose of 250 mg, once a day, everyday. Patients continue treatment until disease progression or unacceptable toxicity. Two dose reductions, 225mg and 150mg, are allowed (200mg and 150mg for patients with a body surface area under 1.65m2) and interruptions of therapy up to two weeks are permitted for recovery from toxicity or intercurrent illness.
Period: Overall Study
Arm/Group | ENMD-2076
Started | 40
Completed | 38
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Of the 40 participants accrued onto trial, 38 were evaluable. Two participants did not complete therapy, and were deemed unevaluable
Groups:
- ENMD-2076: ENMD-2067 will be taken orally at a dose of 275 mg, once a day, everyday for 28 day cycles. Patients with a body surface area of less than 1.65 m2 will receive a starting dose of 250 mg, once a day, everyday for 28 day cycles. Patients can continue on therapy until disease progression or unacceptable toxicity. Dose reductions to 225mg and 150mg (200mg and 150mg for patients with body surface under 1.65m2) are permitted, with up to two weeks of therapy interruptions permitted for recovery from toxicity or intercurrent illness.
Arm/Group | ENMD-2076
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 54 [39 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Prior Therapy [Count of Participants; unit: Participants]
  1 previous therapy | 22
  2 previous therapies | 12
  3 previous therapies | 4

OUTCOME MEASURES:

1. Primary Outcome: Six Month Progression Free Survival Rate
Description: Progression Free Survival (PFS) is defined as the time from first day of treatment to the first observation of disease progression or death due to any cause or last follow up. PFS will be censored for patients who are alive and free of progression at time of last follow-up.
Time Frame: Response will be determined based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1. Progression free survival is the time from the first day of treatment to the first observation of disease progression or Death/last F/U.
Population: Of the 40 participants enrolled, 38 were deemed eligible for evaluation. Two patients did not complete one cycle of therapy and were considered not evaluable.
Measure: Count of Participants; unit: Participants
Groups:
- ENMD-2076: ENMD-2067 will be taken orally at a dose of 275 mg, once a day, everyday. Patients with a body surface area of less than 1.65 m2 will receive a starting dose of 250 mg, once a day, everyday. Patients will continue on therapy until disease progression or unacceptable toxicity. Dose reductions to 225mg and 150mg (200mg and 150mg for patients with body surface area under 1.65m2) are permitted, along with up to two weeks of therapy interruption for recovery from toxicity or intercurrent illness.
Arm/Group | ENMD-2076
Number analyzed (Participants) | 38
Participants | 8

2. Primary Outcome: Complete or Partial Response Rate
Description: Percentage of patients with complete or partial response as per RECIST 1.1 criteria.
Time Frame: 2 years
Population: Of the 40 participants enrolled onto trial, 38 were deemed eligible for evaluation. 2 patients did not complete a cycle of therapy and were considered ineligible for evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- ENMD-2076: ENMD-2067 will be taken orally at a dose of 275 mg, once a day, everyday. Patients with a body surface area of less than 1.65 m2 will receive a starting dose of 250 mg, once a day, everyday. Patients will continue therapy until disease progression or unacceptable toxicity. Dose reductions to 225mg and 150mg (200mg and 150mg for patients with body surface area under 1.65m2) are permitted, along with up to two weeks of interrupted therapy for recovery from toxicities or intercurrent illness.
Arm/Group | ENMD-2076
Number analyzed (Participants) | 38
Participants | 3

3. Secondary Outcome: Time to Disease Progression
Description: Length of time until disease progression in patients treated with ENMD-2076
Time Frame: 2 years
Population: Data not collected.
Arm/Group | ENMD-2076
Number analyzed (Participants) | 0

4. Secondary Outcome: Levels of Certain Proteins and Gene Expression Compared to Patient Outcome Following Treatment
Description: Association of somatic mutations in PIK3CA, ARID1A and PTEN mutation status, and ARID1A and PTEN expression assessed in archival samples and tumour biopsies with tumour response and patient outcome following treatment with ENMD 2076.
Time Frame: 2 years
Population: Data not collected
Arm/Group | ENMD-2076
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All AEs will be recorded in the source documents. All AEs, including clinically significant abnormal laboratory AEs, will be entered in the electronic CRFs from the time of the first dose of study medication until up to 30 days after the end of study drug administration or until alternate therapy is initiated, whichever occurs first.
Arm/Group | ENMD-2076
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 10/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENMD-2076 (N=40)
Hypertension (Cardiac disorders) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Confusion (Psychiatric disorders) | 2 (2)
Vaginal Fistula (Reproductive system and breast disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea & Vomiting (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Dyaphagia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENMD-2076 (N=40)
Fatigue (General disorders) | 28 (28)
Nausea (Gastrointestinal disorders) | 27 (27)
Constipation (Gastrointestinal disorders) | 23 (23)
Diarrhea (Gastrointestinal disorders) | 20 (20)
Hypomagnesemia (Metabolism and nutrition disorders) | 19 (19)
Headache (General disorders) | 18 (18)
Vomiting (Gastrointestinal disorders) | 16 (16)
Weight Loss (General disorders) | 15 (15)
Hypoalbuminemia (Blood and lymphatic system disorders) | 15 (15)
Proteinuria (Renal and urinary disorders) | 14 (14)
Anemia (Blood and lymphatic system disorders) | 13 (13)
Alkaline Phosphatase Increase (Blood and lymphatic system disorders) | 11 (11)
Palmar-Plantar Erythrodysesthensia (Skin and subcutaneous tissue disorders) | 10 (10)
Dysguesia (Nervous system disorders) | 10 (10)
White Blood Cell Decrease (Blood and lymphatic system disorders) | 9 (9)
Dizziness (Nervous system disorders) | 9 (9)
Hypocalcemia (Blood and lymphatic system disorders) | 9 (9)
Elevated TSH (Endocrine disorders) | 9 (9)
Hypothyroidism (Endocrine disorders) | 8 (8)
Mucositis (General disorders) | 8 (8)
AST Increased (Blood and lymphatic system disorders) | 7 (7)
Hypophosphatemia (Blood and lymphatic system disorders) | 6 (6)
ALT Increased (Blood and lymphatic system disorders) | 6 (6)
Hyponatremia (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes